CLINICAL TRIAL: NCT07049458
Title: A Phase I/IIa, Open-Label, Dose-Escalation and Cohort-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CHO-A04 in Subjects With Advanced Solid Tumors
Brief Title: Study of CHO-A04 in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cho Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHO-A04-001
Record Dates: First submitted 2025-06-05; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumor; Anti-SSEA-4 antibody; Monoclonal antibody; Dose-escalation

STUDY DESIGN:
Intervention Model Description: * Phase I: accelerated titration and traditional 3+3 dose-escalation design
  * Phase II: cohort-expansion design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase I Dose Level -1: 0.5 mg/kg/week (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase I Dose Level 1: 1 mg/kg/week [starting dose] (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase I Dose Level 2: 2 mg/kg/week (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase I Dose Level 3: 4 mg/kg/week (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase I Dose Level 4: 8 mg/kg/week (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase I Dose Level 5: 12 mg/kg/week (Experimental): Intravenous infusion weekly
  Interventions: Drug: CHO-A04
- Phase IIa: RP2D for Cancer type A (Experimental): Recommended Phase II dose (RP2D) level will be decided by Scientific Review Committee (SRC) based on accumulated study data in Phase I. Cancer type of each cohort will be determined before initiation of Phase IIa
  Interventions: Drug: CHO-A04
- Phase IIa: RP2D for Cancer type B (Experimental): Recommended Phase II dose (RP2D) level will be decided by Scientific Review Committee (SRC) based on accumulated study data in Phase I. Cancer type of each cohort will be determined before initiation of Phase IIa
  Interventions: Drug: CHO-A04

INTERVENTIONS:
Drug: CHO-A04 — CHO-A04 will be given intravenously (IV) once weekly for 4 weeks as a treatment cycle.

SUMMARY:
The goal of this clinical trial is to learn if the study drug, CHO-A04, works to treat solid cancers in adults. It will also aim to learn about the safety of CHO-A04 and find the best dose to use in future cancer treatment. The main questions it aims to answer are:

* Which dose of CHO-A04 shows the best anti-cancer ability?
* How will your body respond to CHO-A04 treatment?
* How long will CHO-A04 remain in your body?

There are two stages of investigation in this study:

* Phase I: to find the best anti-cancer dose of CHO-A04
* Phase IIa: to find the CHO-A04 anti-cancer ability in specific cancer types

In this study, each participant will be assigned to one of the CHO-A04 dose levels. Participants will have CHO-A04 infusion via blood vessel once every week for four weeks. The CHO-A04 treatment may continue based on participants' condition and CHO-A04 safety evaluations.

DETAILED DESCRIPTION:
This Phase I/IIa, open-label, dose-escalation and cohort-expansion study aims to evaluate the safety, pharmacokinetics, and preliminary efficacy of CHO-A04 in subjects aged ≥ 18 years with advanced solid tumors.

Both Phases I and Phase IIa include a screening period of up to 4 weeks and study treatment once every week starting from Cycle 1 Day 1 (C1D1) until any treatment discontinuation criterion is met. Each treatment cycle of the study treatment is 28 days.

Subjects will receive intravenous (IV) infusion of CHO-A04 once a week for 4 weeks (D1, D8, D15, D22) as a treatment cycle. After the completion of last dose of the study treatment, subjects should complete the end-of-treatment (EOT) visit, safety follow-up (EOS) visit, and survival follow-up visits, unless withdrawn from this study.

- Phase I (accelerated titration and traditional 3+3 dose-escalation): Phase I consists of the accelerated titration and the traditional 3+3 dose-escalation design. Eligible subjects will be sequentially assigned into one of the dose levels. Dose level will be escalated from dose level 1 (starting dose) at 1 mg/kg/week to dose level 5 at 12 mg/kg/week of CHO-A04 (or may be de-escalated to dose level -1 at 0.5 mg/kg/week). If any ≥ Grade 2 CHO-A04 related adverse events (AEs) occurs in dose level 1 or dose level 2 subjects, the dose escalation/de-escalation rule will follow the 3+3 design. Intra-subject dose-escalation is not allowed in this study.

- Phase IIa (cohort-expansion): Two cohorts of up to 10 subjects per cohort will receive the Recommend Phase 2 Dose (R2PD), which is a dose equal to or lower than MTD based on the SRC's decision. The Sponsor will determine the cancer type for each cohort before initiation of Phase IIa.

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged ≥ 18 years
2. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors
3. Must have been treated with established standard-of-care therapy, or physicians have determined that such established therapy is not sufficiently efficacious, or patients have declined to receive standard-of-care therapy
4. Availability of archival tissue specimens for SSEA-4 immunohistochemistry (IHC) staining (optional for Phase I). Acceptable tumor tissues include:

   1. Tumor tissue sample collected at the time of initial diagnosis
   2. The most recent available recurrent/metastatic tumor biopsy tissue is preferred if available (a pre-treatment biopsy is encouraged if the biopsy site is safely accessible) Note: This criterion is fulfilled if there is a qualified tumor sample (tumor cells were presented in the tumor biopsy tissue) and the tumor tissue slides can be obtained for IHC staining. It is not violated even if the staining result obtained after the screening visit reveals that the slides contain no identifiable tumor cells.
5. Has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
7. Has a life expectancy of at least 12 weeks in the opinion of the Investigator
8. Has adequate hematopoietic function:

   1. Absolute neutrophil count (ANC) ≥ 1500 cells/μL without the need of myeloid growth factor support within 1 week
   2. Platelet ≥ 90×103 counts/μL without the need of platelet transfusion support within 1 week
   3. Hemoglobin ≥ 9.0 g/dL without the need of red blood cell (RBC) transfusion within 1 week
9. Has adequate coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5× upper limit of the normal range (ULN)
10. Has adequate liver function:

    1. Total bilirubin ≤ 1.5× ULN and no signs of jaundice (≤ 3× ULN for subjects with known Gilbert disease)
    2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN or ≤ 5.0× ULN in case of documented hepatic metastasis or hepatocellular carcinoma (HCC). For subjects with HCC, the Child-Pugh score must be ≤ 6
11. Has adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2) Note: eGFR (mL/min/1.73 m2) = 186.3 × (serum creatinine in mg/dL)-1.154 × (age)-0.203× (0.742 if female) × (1.212 if African American/black)
12. Willingness and ability to comply with protocol-stated requirements, instructions, and restrictions per Investigator's judgment
13. Is able to understand the nature of this clinical study and accepts to enter the study by signing the informed consent form (ICF)

Exclusion Criteria:

1. Has unresolved toxicities from prior anticancer therapy, defined as having not resolved to ≤ Grade 1 (NCI-CTCAE v5.0), except for alopecia and laboratory values listed in the inclusion criteria
2. Has signs or symptoms of end-stage organ failure, major chronic illnesses other than cancer(s), or any severe concomitant conditions which, in the Investigator's opinion, make it undesirable for the subject to participate in the study, or could jeopardize compliance with the protocol
3. History of another primary malignancy within the last 3 years (except for treated basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, or in situ cancer of the cervix) prior to the planned first infusion
4. Has any significant cardiovascular or pulmonary diseases, including:

   1. Poorly controlled hypertension (systolic blood pressure ≥ 160 mm Hg and diastolic blood pressure ≥ 100 mm Hg)
   2. Left ventricular ejection fraction (LVEF) < 50% at the screening visit
   3. Congestive heart failure (defined as New York Heart Association Class III or IV), myocarditis, myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, or coronary artery bypass graft within 24 weeks prior to the planned first infusion
   4. Uncontrolled serious cardiac arrhythmias, such as ongoing clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation or Torsades de Pointes) Note: Sustained ventricular tachycardia is defined as tachycardia that continues for more than 30 seconds or leads to hemodynamic compromise within 30 seconds and requires intervention
   5. Corrected QT interval (QTcF) > 480 ms demonstrated by at least two 12-lead ECGs > 30 minutes apart
   6. Evidence of active pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or history of idiopathic pulmonary fibrosis. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
   7. History of 2nd or 3rd-degree atrioventricular conduction defects
5. History of thromboembolic or cerebrovascular events within the last 24 weeks before the screening visit, including transient ischemic attack, cerebrovascular accident, or deep vein thrombosis
6. Has other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would make the subject inappropriate for enrollment in this study in the opinion of the Investigator
7. Has received anti-cancer therapies such as surgery on target lesions, chemotherapy, small molecule agent(s), hormone therapy, radiation therapy (except for palliative radiotherapy for bone metastasis of non-skeletal tumors), or any other anti-cancer agent(s) within 4 weeks or 5 half-lives of the treated agents, whichever is longer, prior to the first dosing. Has received prior anti-cancer monoclonal antibody therapy within 8 weeks prior to the first infusion.
8. Has received systemic immunosuppressive medication(s) (including, but not limited to, steroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, tumor necrosis factor-ɑ antagonists, and calcineurin inhibitors) within 2 weeks (for those with a half-life ≤ 72 hours) or 4 weeks (for those half-life > 72 hours) prior to study dosing.

   Note: For regular steroid use, ≤ 10 mg of prednisolone per day or equivalent is allowed. Inhaled or topical corticosteroids are allowed.
9. Has participated in other clinical studies for investigational product(s) or medical device within 4 weeks or 5 half-lives (if known) prior to the planned first infusion, whichever is longer
10. Has received cell therapy within 12 weeks prior to the planned first infusion
11. Prior allogeneic hematopoietic stem cell, solid organ, or bone marrow transplantation(s)
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

    Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the planned first infusion and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases. This exception does not include carcinomatous meningitis which is excluded regardless of its clinical stability
13. Has symptomatic or poorly controlled pleural effusion, pericardial effusion, or ascites
14. With the following infections:

    1. History of active pulmonary tuberculosis infection ≤ 48 weeks prior to the planned first infusion, regardless of tuberculosis treatment
    2. Any major episode of infection requiring treatment with systemic antibiotics or hospitalization within 4 weeks prior to the planned first infusion
    3. Positive HBsAg; subjects with positive HBsAg test results can be considered as eligible if subjects can receive anti-HBV viral treatment(s), e.g., entecavir or tenofovir
    4. Positive anti-HCV; subjects with positive for anti-HCV but with negative results for HCV viremia as shown by PCR are considered as eligible.
    5. Medical history showing confirmed HIV-1 positivity
15. Administration of a live, attenuated vaccine within 4 weeks prior to the planned first infusion or anticipation that such a live, attenuated vaccine will be required during the treatment period.
16. With known or suspected hypersensitivity to any ingredients of investigational product
17. History of severe allergic, anaphylactic, or other severe hypersensitivity reactions to therapeutic humanized antibodies
18. Female subject who is breastfeeding, has a positive pregnancy test result at eligibility checking, or expecting to conceive or have children within the projected duration of the trial, starting from the screening visit through 90 days after the last dose of study treatment.
19. All male subjects and female subjects with childbearing potential* (between puberty and 2 years after menopause) refuse to use at least two of appropriate contraception methods shown below from signing the ICF to at least 3 months after taking the last dose of study treatment.

    1. Use oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

       * Male or female subjects who have undergone the following procedures are considered without childbearing potential.

         * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 12 weeks before the screening visit. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
         * Male sterilization (24 weeks prior to the first infusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with dose-limiting toxicity (DLT) | Up to 28 days after first dose (Cycle 1)
  DLT is evaluated based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.The 5 general grades includes Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening or disabling, and Grade 5: Death.
Percentage of subjects occur with adverse events (AEs) | Up to 30 days after the last dose
  Percentage of subjects with treatment-emergent adverse events (TEAEs), treatment-related adverse event (TRAEs), serious adverse events (SAEs), and infusion-related reactions (IRRs) will be measured. Severity grading will be assessed by the investigator based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. The 5 general grades includes Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening or disabling, and Grade 5: Death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From first dose to disease progression or death, whichever occurs first, assessed up to 12 months
  Progression-free survival (PFS) is defined as the time from the date of initial dosing until the first date of either disease progression or death due to any cause.
Overall response rate (ORR) | CT assessment every 2 cycles throughout the study till EOT follow-up
  ORR will be calculated by combining subjects with complete response (CR) or partial response (PR) based on RECIST v1.1 criteria in best response.
Disease control rate (DCR) | From first dose to confirmed disease progression, assessed up to 12 months
  DCR is defined as the percentage of subjects with at least one complete response (CR), partial response (PR) or stable disease (SD) per RECIST v1.1.
Duration of response (DOR) | From date of first documented response (CR or PR) to date of disease progression or death, assessed up to 12 months
  DOR is defined as time from the date of the first documentation of partial response (PR) or complete response (CR) per RECIST v1.1 to the date of progression
Change in Eastern Cooperative Oncology Group (ECOG) performance score from baseline | Throughout the study till 4 weeks after the last dose
  ECOG performance status is a scale used to assess how the disease affects the daily living abilities, and determine appropriate treatment and prognosis. It is a simple measure of functional status that determines ability of patient to tolerate therapies in cancer. The grading ranges from 0 (fully active, without performance restriction) to 5 (dead).
Blood Concentration of CHO-A04 | From day 1 pre-dosing, various time point after dosing and throughout the study till EOT follow-up (assessed up to 12 months)
  The concentration of CHO-A04 in blood
Anti-drug antibodies (ADAs) concentration | Baseline, various time point during treatment period, and EOT follow-up (assessed up to 12 months)
  The concentration of ADA in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi (Josh) Lin, M.D., PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No